CLINICAL TRIAL: NCT03333200
Title: Longitudinal Study of Neurodegenerative Disorders
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Deepa Soundara Rajan, Associate Professor, University of Pittsburgh
Other Study IDs: STUDY19020318
Record Dates: First submitted 2017-04-24; First posted 2017-11-06 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: MLD; Krabbe Disease; ALD; MPS I; MPS II; MPS III; Vanishing White Matter Disease; GM3 Gangliosidosis; PKAN; Tay-Sachs Disease; NP Deficiency; Osteopetrosis; Alpha-Mannosidosis; Sandhoff Disease; Niemann-Pick Diseases; MPS IV; Gaucher Disease; GAN; GM1 Gangliosidoses; Morquio Disease; S-Adenosylhomocysteine Hydrolase Deficiency; Batten Disease; Pelizaeus-Merzbacher Disease; Leukodystrophy; Lysosomal Storage Diseases; Purine Nucleoside Phosphorylase Deficiency; Multiple Sulfatase Deficiency Disease
Keywords: Pediatric; Rare; Neurodegenerative; Genetic; Neurodevelopment; Brain; MRI; Biorepository; NDRD; Longitudinal; Cognitive; Motor; Language; Adaptive behavior
MeSH Terms: conditions — Leukodystrophy, Globoid Cell; Sudden Infant Death; Mucopolysaccharidosis III; Leukoencephalopathies; Tay-Sachs Disease; Purine Nucleoside Phosphorylase Deficiency; Osteopetrosis; alpha-Mannosidosis; Sandhoff Disease; Niemann-Pick Diseases; Mucopolysaccharidosis IV; Gaucher Disease; Hypermethioninemia; Neuronal Ceroid-Lipofuscinoses; Pelizaeus-Merzbacher Disease; Lysosomal Storage Diseases; Multiple Sulfatase Deficiency Disease; Language | interventions — Palliative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — NDRD Biorepository includes: blood plasma and serum, CSF, brain and other tissues
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Palliative Care — Collecting information about the natural progression of these diseases
Biological: Hematopoetic Stem Cell Transplantation — Following patients who have received HSCT as part of their clinical care.

SUMMARY:
The purpose of this study is to understand the course of rare genetic disorders that affect the brain. This data is being analyzed to gain a better understanding of the progression of the rare neurodegenerative disorders and the effects of interventions.

DETAILED DESCRIPTION:
Patients would be evaluated by a multidisciplinary team at specific time points every 3 months the first year, every 6 months the second year and once a year thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a genetic neurodegenerative disorder

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Persons with genetic neurodegenerative diseases.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2012-01-11 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2035-01 (Estimated)

PRIMARY OUTCOMES:
Cognitive development | 15 years
  Repeated standardized age equivalent scores.
Language development | 15 years
  Repeated standardized age equivalent scores.
Gross Motor development . | 15 years
  Repeated standardized age equivalent scores.
Fine Motor development | 15 years
  Repeated standardized age equivalent scores.
Adaptive living skills | 15 years
  Repeated standardized age equivalent scores.

SECONDARY OUTCOMES:
Exploratory biomarkers | 15 years
  Blood, CSF and urine
Neurodegeneration of the brain as measured by MRI diffusion tensor imaging from birth to 5 years of age | 5 years
  Specialized technique to use DTI data to measure brain degeneration over time

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
The IPD will be shared after review and only under a DTA, CDA through our office of research.